CLINICAL TRIAL: NCT02252341
Title: Effects of N-Acetyl-Cysteine on Oxidative Stress Biomarkers in Bipolar Patients With and Without Tobacco Use Disorder
Brief Title: Efficacy of N-Acetyl-Cysteine in Bipolar Disorder and Tobacco Use Disorder
Acronym: NACBD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade Estadual de Maringá (Other)
Responsible Party: Principal Investigator, Mauro Porcu, Professor of Psychiatry, Universidade Estadual de Maringá
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-007
Record Dates: First submitted 2014-07-04; First posted 2014-09-30 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Bipolar Disorder
Keywords: smoking; inflammation; oxidative stress; NAC; treatment
MeSH Terms: conditions — Bipolar Disorder; Smoking; Inflammation | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Dietary Supplement: N-Acetyl-Cysteine Phase 4 Study Type: Interventional Study Design: Treatment, Parallel Assignment, Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor), Randomized, Efficacy Study
  Primary Outcome Measure:
  Hamilton Depression Rating Scale [Time Frame: baseline, 1, 2, 3 months] [Designated as safety issue: Yes]
  Secondary Outcome Measures:
  Carbon Oxide exhalation [Time Frame: basal, 1, 2, 3 months] [Designated as safety issue: Yes]
  Other Pre-specified Outcome Measures:
  Biological outcome measures [Time Frame: baseline and 3 months] [Designated as safety issue: Yes] inflammatory and oxidative stress biomarkers N-Acetyl-cysteine 1800 mg / day will be taken for 12 weeks versus placebo 12 weeks.
- N-Acetyl-Cysteine (Placebo Comparator): Study Type: Interventional Study Design: Treatment, Parallel Assignment, Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor), Randomized, Efficacy Study
  Official Title: Effects of N-Acetyl-Cysteine on Oxidative Stress Biomarkers in Bipolar Patients With and Without Tobacco Use Disorder
  Primary Outcome Measure:
  Hamilton Depression Rating Scale [Time Frame: baseline] [Designated as safety issue: Yes]
  Secondary Outcome Measures:
  Carbon Oxide exhalation [Time Frame: basal, 1, 2, 3 months] [Designated as safety issue: Yes]
  Other Pre-specified Outcome Measures:
  Biological outcome measures [Time Frame: baseline and 3 months] [Designated as safety issue: Yes] inflammatory and oxidative stress biomarkers
  Placebo will be taken for 12 weeks.
  Interventions: Dietary Supplement: N-Acetyl-Cysteine

INTERVENTIONS:
Dietary Supplement: N-Acetyl-Cysteine — drug: N-Acetyl-cysteine N-Acetyl-cysteine 1800 mg a day for 12 weeks versus placebo for 12 weeks
  Other Names: N-acetyl-cysteine 1800 mg a day for 12 weeks or; N-Acetyl-cysteine 3 pills/day for 12 weeks.
  Arms: N-Acetyl-Cysteine

SUMMARY:
Effects of N-Acetyl-Cysteine in patients with bipolar depression (primary outcome is Hamilton Depression Rating Scale) with and without tobacco use disorder and on inflammatory and oxidative stress biomarkers

DETAILED DESCRIPTION:
The study subjects are bipolar depressive patients seeking outpatient treatment for bipolar affective disorder in the psychiatric outpatient clinic in Heath Unit System of the Network of Outpatient Hospital of the State University of Londrina , and tobacco use disorder according of criteria Diagnostic Statistical Manual for Mental Disorders, as control use never smokers.

This is a placebo-controlled, 12 weeks, with a sample of 130 bipolar patients who sought treatment at the outpatient clinic of the Hospital of clinical psychiatry at State University of Londrina clinical trial , double-blind , randomized, from May 2015 to May 2016. Patients will be randomly allocated into two groups, double-blind, to receive a combination product (NAC, 1.8 g/day) or placebo for a period of 12 weeks. Both groups remain receiving maintenance treatment in outpatient psychiatry , and general medical and routinely reviews psychiatric . The dosage will be fixed 1.8 g /day of NAC administered in capsules taken 1 before breakfast, 1 before lunch and 1 before dinner is equal doses.

The choice of this dosage is based on previous studies (Prado et al., submitted) , in which similar doses that are effective and well tolerated . To enable the process to be double-blind study medications (NAC or placebo ) will be dispensed monthly number and identical formulations and packages sealed by a pharmacist who will participate in the parallel test . Patients will do blood tests for assessment of oxidative stress at baseline will be randomized to use of NAC or placebo and at the final stage of the 12 weeks , when the new assessment and collection of blood for analysis of oxidative stress will be performed . Clinicians who conduct the study will be blinded to allocation of NAC or placebo for each patient .

The NAC is a compound with a low rate of adverse effects , among them being described diarrhea, nausea and dermatological allergy. It is considered a very low risk medication. The placebo will be the basis of lactose, composed almost devoid of risk for side effects except if allergic to lactose (exclusion criterion ) .

ELIGIBILITY:
Inclusion Criteria:

To be included in this study participants between 18 and 65 years, both sexes , all races, capacity to consent to the study and carefully follow the guidelines and procedures and sign the term of free and informed consent. Patients with bipolar depression will be included with score above 21 on the Hamilton Depression Rating Scale (17 items) and above 14 on the Beck Depression Inventory.

Exclusion Criteria:

We will exclude: patients with delirium or cognitive deficits or failure of understanding and reflection to change. Furthermore, dementia , amnesia and other cognitive disorders, infectious diseases such as hepatitis B and C , HIV, chronic diseases such as renal failure, obstructive pulmonary disease and autoimmune interferon treatment, stroke , Parkinson's disease, pathological use of psychoactive substances and consumption of antioxidants. These situations can affect an inflammatory and / or immune process

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
number cigarettes per day | baseline

SECONDARY OUTCOMES:
Carbon Oxide exhalation | basal, 1, 2 and 3 months

OTHER OUTCOMES:
Biological outcome measures | baseline and 3 months
  inflammatory and oxidative stress biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Nunes, M.D, Ph.D, Study Chair — Universidade Estadual de Londrina
Locations (1):
- State University of Maringá, Maringá, Paraná, Brazil

REFERENCES:
- [Derived] Porcu M, Urbano MR, Verri WA Jr, Barbosa DS, Baracat M, Vargas HO, Machado RCBR, Pescim RR, Nunes SOV. Effects of adjunctive N-acetylcysteine on depressive symptoms: Modulation by baseline high-sensitivity C-reactive protein. Psychiatry Res. 2018 May;263:268-274. doi: 10.1016/j.psychres.2018.02.056. Epub 2018 Mar 13. PMID 29605103
- See also: departement of medicine - state university of Maringá — http://www.dmd.uem.br